CLINICAL TRIAL: NCT00588731
Title: Cannabinoid Receptor Antagonist Treatment of Cognitive Dysfunction in Schizophrenia
Brief Title: Cannabidiol Treatment of Cognitive Dysfunction in Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Mohini Ranganathan, Assistant Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0710003164; 07TGS-1082
Record Dates: First submitted 2007-12-29; First posted 2008-01-09 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cannabidiol (Experimental)
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — Active Cannabidiol daily over 6 weeks
  Arms: Cannabidiol
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is a six-week, randomized, placebo-controlled, fixed dose trial comparing cannabidiol Vs. placebo added to a stable dose of antipsychotic medications in patients diagnosed with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia or Schizoaffective disorder (DSM-IV SCID-confirmed),

Exclusion Criteria:

* Women who are pregnant, nursing or unwilling to use appropriate birth control measures during study participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohini Ranganathan, M.D., Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Boggs DL, Surti T, Gupta A, Gupta S, Niciu M, Pittman B, Schnakenberg Martin AM, Thurnauer H, Davies A, D'Souza DC, Ranganathan M. The effects of cannabidiol (CBD) on cognition and symptoms in outpatients with chronic schizophrenia a randomized placebo controlled trial. Psychopharmacology (Berl). 2018 Jul;235(7):1923-1932. doi: 10.1007/s00213-018-4885-9. Epub 2018 Apr 5. PMID 29619533

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cannabidiol | Placebo
Started | 21 | 20
Completed | 18 | 18
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Population: A total of 36 participants completed all aspects of the study. Higher T-scores represent better outcomes.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cannabidiol | Placebo | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (9.3) | 46.4 (9.5) | 47.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 12 | 13 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 12 | 19
  White | 10 | 5 | 15
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36
Length of Diagnosis [Mean (Standard Deviation); unit: years] | 25.6 (12.7) | 28.2 (8.5) | 26.9 (10.6)
Intelligence Quotient (IQ) [Mean (Standard Deviation); unit: IQ] | 91.6 (18.4) | 82.3 (15.4) | 86.6 (17.3)
Education [Mean (Standard Deviation); unit: years] | 13.2 (1.6) | 12.8 (2) | 13 (1.8)
Smoking Status [Number; unit: participants]
  Smokers | 9 | 10 | 19
  Non-Smokers | 9 | 8 | 17
Hopkins Verbal Learning Test T-Score [Mean (Standard Deviation); unit: T-Score] — The Hopkins Verbal Learning Test is a measure of verbal short term memory. Each trial has a max total score of 12 (range of 0-12), and the max total score for all three trials is 36 (range of 0-36). The data listed is reported in the form of a t-score, with a higher score representing better verbal learning. These t-score values are normalizing the scores to populations, comparing them to a representative sample.
  T-Score | 32.5 (6.3) | 34.5 (6) | 33.5 (6.15)
Positive And Negative Syndrome Scale [Mean (Standard Deviation); unit: T-score] — The PANSS is a scale used for measuring symptoms severity of patients with schizophrenia. Of the 30 items included: 7 constitute a Positive Scale, 7 a Negative Scale, and 16 a General Psychopathology Scale. The scores for these scales are arrived at by summation of ratings across component items (each item scored between 1-7). Therefore, the potential ranges are 7-49 for the Positive and Negative Scales, and 16-112 for the General Psychopathology Scale. The PANSS Total Score is the summation of these subscales and can range from a score of 30-210. A higher score indicates more severe symptoms.
  T-score
    PANSS Total Score | 76.6 (17) | 82.7 (8.8) | 79.65 (12.9)
    PANSS Positive Subscale | 18.8 (4.7) | 20.6 (3.8) | 19.7 (4.25)
    PANSS Negative Subscale | 20.7 (4.6) | 20.9 (4.7) | 20.8 (4.65)
    PANSS General Subscale | 37.1 (10.3) | 41.2 (5.6) | 39.15 (7.95)
Medications [Number; unit: participants]
  First Generation Antipsychotics | 9 | 5 | 14
  Second Generation Antipsychotics | 10 | 13 | 23
  Multiple Antipsychotics | 2 | 7 | 9
  Long Acting Injectable Antipsychotics | 3 | 6 | 9
  Antidepressant | 3 | 4 | 7
  Anticholinergic | 7 | 7 | 14
  Anticonvulsants/Mood Stabilizers | 3 | 6 | 9
  Benzodiazepine | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Verbal Short Term Memory
Description: Verbal short term memory is measured through the Hopkins Verbal Learning Test. Each trial has a max total score of 12 (range of 0-12), and the max total score for all three trials is 36 (range of 0-36). However, the data listed below is reported in the form of a t-score, with a higher score representing better verbal learning. These t-score values are normalizing the scores to populations, comparing them to a representative sample, with a mean of 50.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Cannabidiol | Placebo
Number analyzed (Participants) | 18 | 18
t-score
  Baseline | 43.7 (9.7) | 37.9 (7.4)
  Endpoint | 43.6 (10.8) | 40.8 (8.5)
Statistical Analysis 1: Comparison: Cannabidiol vs Placebo; Test type: Superiority or Other; p = 0.90, ANOVA

2. Secondary Outcome: Overall Cognition as Measured on the MATRICS Battery
Description: Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) is intended to provide a relatively brief evaluation of key cognitive domains relevant to schizophrenia and related disorders. A higher score indicates better cognition (i.e. speed of processing, attention, verbal and non-verbal working memory, visual learning, reasoning, problem solving, and social cognition). The below scores are t-score values, which are normalized scores to the population and comparing the scores to a representative sample.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | Cannabidiol | Placebo
Number analyzed (Participants) | 18 | 18
t-score
  Baseline | 27.8 (14) | 23.2 (13.3)
  Endpoint | 26.4 (12.2) | 25.4 (12.5)
Statistical Analysis 1: Comparison: Cannabidiol vs Placebo; Test type: Superiority or Other; p = 0.76, ANOVA

ADVERSE EVENTS:
Arm/Group | Cannabidiol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 15/21 | 17/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cannabidiol (N=21) | Placebo (N=20)
Social Stress (Social circumstances) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Appetite Changes (Metabolism and nutrition disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 4
Abnormal Dreams (Psychiatric disorders) | 1 | 2
Dry Mouth (Gastrointestinal disorders) | 3 | 2
Endocrine (Endocrine disorders) | 1 | 1
Extrapyramidal Side Effects (Nervous system disorders) | 1 | 0
Feeling "High" (Psychiatric disorders) | 1 | 0
Gastrointestinal (Gastrointestinal disorders) | 6 | 10
Infection (Infections and infestations) | 4 | 4
Pain (Nervous system disorders) | 7 | 7
Photosensitivity (Eye disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Salivation (Gastrointestinal disorders) | 0 | 1
Sedation (Nervous system disorders) | 4 | 1
Sexual Side Effects (Reproductive system and breast disorders) | 1 | 2
Sleep (Nervous system disorders) | 2 | 5
Taste (Gastrointestinal disorders) | 0 | 1
Tension (Psychiatric disorders) | 0 | 1
Visual Changes (Psychiatric disorders) | 0 | 1
Weight Change (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No